CLINICAL TRIAL: NCT07325331
Title: Effects of Lullaby, White Noise, and Silent Headphone Use on Sedation Depth, Anesthetic Requirements, and Recovery Time in Children Undergoing MRI: A Prospective Randomized Controlled Trial
Brief Title: Lullaby vs White Noise vs Silence in Pediatric MRI Sedation
Acronym: CALMMRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil,MD, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 12.2.2025-
Record Dates: First submitted 2025-12-02; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Sedation

STUDY DESIGN:
Intervention Model Description: Three-arm, parallel-group, randomized controlled design evaluating the effects of lullaby music, white noise, and silent headphone use on sedation depth, anesthetic requirements, and recovery outcomes during pediatric MRI
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcome assessors are blinded to group allocation. Only the radiology technician operating the MRI scanner and initiating the auditory condition (lullaby, white noise, or silent headphones) is aware of the assignment; the technician is not involved in sedation management or outcome assessment."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silent Headphone Group (Other): Participants wear MRI-compatible headphones without any auditory input. No music or noise is delivered throughout the MRI procedure. Standard sedoanalgesia is administered according to institutional protocol.
  Interventions: Behavioral: Silent Headphone
- White Noise Group (Other): Participants receive continuous white noise through MRI-compatible headphones starting immediately after sedoanalgesia and continuing throughout the MRI examination. All other clinical care follows standard pediatric sedation practice.
  Interventions: Behavioral: White Noise
- Lullaby Music Group (Other): Participants receive continuous lullaby music through MRI-compatible headphones beginning after sedoanalgesia and continuing for the duration of the MRI procedure. Sedation and monitoring follow standard institutional protocols.
  Interventions: Behavioral: Lullaby Music

INTERVENTIONS:
Behavioral: Silent Headphone — Use of MRI-compatible headphones without auditory input during the MRI procedure.
  Arms: Silent Headphone Group
Behavioral: White Noise — Continuous delivery of white noise through MRI-compatible headphones throughout the MRI procedure
  Arms: White Noise Group
Behavioral: Lullaby Music — Continuous delivery of lullaby music through MRI-compatible headphones for the duration of the MRI examination
  Arms: Lullaby Music Group

SUMMARY:
This prospective randomized study aims to evaluate the effects of three auditory conditions-lullaby music, white noise, and silent headphone use-on sedation depth, anesthetic drug requirements, and recovery outcomes in children undergoing MRI. A total of 150 pediatric patients aged 6 months to 12 years will be assigned to one of three groups: lullaby, white noise, or silent headphone (isolation) control. All participants will receive routine sedoanalgesia according to institutional protocol. Vital signs, sedation depth, movement requiring sequence repetition, additional anesthetic dosing, and intra-procedural complications will be recorded. Post-procedure recovery will be assessed using the Ramsey Sedation Scale and the Modified Aldrete Score until discharge criteria are met. The study will compare whether auditory stimulation influences sedation stability, reduces anesthetic consumption, and improves recovery time during pediatric MRI.

DETAILED DESCRIPTION:
This prospective randomized study is designed to investigate the effects of three auditory conditions-lullaby music, white noise, and silent headphone use-on sedation depth, anesthetic drug requirements, motion-related sequence repetition, and recovery outcomes during pediatric magnetic resonance imaging (MRI). Children aged 6 months to 12 years who require MRI under sedation will be enrolled. Participants will be randomly assigned to one of three groups: (1) silent headphone control, (2) white noise, or (3) lullaby music. Auditory stimulation in the white noise and lullaby groups will begin immediately after sedoanalgesia and will continue uninterrupted throughout the MRI examination. The control group will wear headphones without any auditory input.

Standard sedoanalgesia will be administered according to institutional pediatric anesthesia practice. During the MRI procedure, heart rate, oxygen saturation, and respiratory rate will be monitored continuously, with values recorded at 5-minute intervals. Any movement that compromises image quality will be documented, including the need for additional anesthetic dosing and repetition of imaging sequences. Procedure-related complications will also be recorded.

Following completion of the MRI, all participants will be transferred to the recovery area, where sedation and recovery assessments will be performed using the Ramsey Sedation Scale and the Modified Aldrete Score until discharge criteria are met. Demographic variables, diagnosis, MRI region, contrast use, total sedation time, MRI duration, auditory stimulation duration, anesthetic doses administered before and during MRI, and total time to discharge will be recorded for outcome comparison.

The study aims to determine whether specific auditory stimuli can enhance sedation stability, minimize anesthetic drug requirements, reduce movement-related interruptions, and shorten recovery time in pediatric patients undergoing MRI. The findings may help identify non-pharmacologic strategies to optimize pediatric sedation, improve imaging quality, and enhance patient safety in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 months and 12 years.
* Scheduled to undergo MRI requiring sedation.
* American Society of Anesthesiologists (ASA) Physical Status I-III.
* Able to use MRI-compatible headphones.
* Parent or legal guardian able to provide written informed consent.

Exclusion Criteria:

* Age under 6 months or over 12 years.
* Known allergy, intolerance, or contraindication to sedative medications used in institutional protocols.
* History of airway anomalies, difficult airway, or conditions increasing anesthesia risk.
* Hearing impairment or auditory limitations preventing perception of sound stimuli.
* Contraindications to MRI (e.g., metallic implants, pacemaker, severe claustrophobia).
* Inability to obtain informed consent from parent or legal guardian.
* Sedation failure or unsuccessful MRI procedure.
* Use of medications or medical conditions that may interfere with sedation assessment or auditory perception.
* Acute respiratory infection or active upper airway disease that increases sedation risk

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
Total Anesthetic Drug Consumption | Periprocedural (during MRI examination)
  Total amount of sedative/anesthetic medication administered during the MRI procedure, recorded in milligrams. Includes initial and additional doses required due to movement or inadequate sedation.

SECONDARY OUTCOMES:
Sedation Depth | Immediately at the end of the MRI procedure
  Depth of sedation will be assessed using the Ramsey Sedation Scale immediately following completion of the MRI examination. Higher scores indicate deeper sedation.
Motion Requiring Sequence Repetition | Periprocedural (during MRI examination)
  Number of MRI sequences repeated due to patient movement that compromises image quality. The total count of repeated sequences will be compared among the three auditory intervention groups.
Recovery Time | assessed up to 120 minutes post-procedure
  Time interval from the end of the MRI examination until the patient reaches a Modified Aldrete Score ≥ 9 in the recovery area. This measure reflects post-sedation recovery efficiency
Heart Rate During MRI | Periprocedural (during MRI scan)
  Heart rate will be continuously monitored and recorded at 5-minute intervals throughout the MRI procedure. Heart rate values will be analyzed to assess sedation stability and compared among the three auditory conditions.
Postoperative Nausea | Assessed Periprocedural and up to 120 minutes post-procedure
  Presence or absence of postoperative nausea assessed during the first 24 hours after surgery. The occurrence will be recorded as a binary outcome (yes/no).
Postoperative Vomiting | Assessed Periprocedural and up to 120 minutes post-procedure
  Occurrence of postoperative vomiting during the first 24 hours after surgery. The occurrence will be recorded as a binary outcome (yes/no).
Incidence of Oxygen Desaturation | Assessed Periprocedural and up to 120 minutes post-procedure
  Oxygen desaturation will be defined as a peripheral oxygen saturation (SpO₂) value below 90% lasting for at least 10 seconds during the procedure. The occurrence of oxygen desaturation will be recorded as a binary variable (yes/no) and compared among the three study groups.
Incidence of Airway Obstruction | Assessed Periprocedural and up to 120 minutes post-procedure
  Airway obstruction will be defined as the presence of clinical signs requiring airway intervention, including jaw thrust, chin lift, insertion of an airway adjunct, or bag-mask ventilation. Events will be recorded as present or absent and compared among the three study groups.
Incidence of Unexpected Agitation | Assessed Periprocedural and up to 120 minutes post-procedure
  Unexpected agitation will be defined as agitation requiring additional sedative or anesthetic intervention or interruption of the procedure, corresponding to a Richmond Agitation-Sedation Scale (RASS) score of +2 or higher. The occurrence will be recorded as a binary outcome (yes/no) and compared among the three study groups.
Oxygen Saturation During MRI | Periprocedural (during MRI scan)
  Peripheral oxygen saturation (SpO₂) will be continuously monitored and recorded at 5-minute intervals during the MRI procedure. SpO₂ values will be analyzed to evaluate sedation stability and compared among the three auditory conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Acil, M.D., Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gergin OO, Pehlivan SS, Erkan I, Bayram A, Aksu R, Gorkem SB, Bicer C, Yildiz K. The effect of playing music and mother's voice to children on sedation level and requirement during pediatric magnetic resonance imaging. Explore (NY). 2023 Jul-Aug;19(4):600-606. doi: 10.1016/j.explore.2023.01.001. Epub 2023 Jan 7. PMID 36628804